CLINICAL TRIAL: NCT01867658
Title: A Prospective Multi-Center Clinical Study to Evaluate the Safety of Progel® Pleural Air Leak Sealant in Video Assisted and Robotic Assisted Thoracotomy Surgery
Brief Title: Progel® Pleural Air Leak Sealant (PALS) in Video and Robotic Assisted Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO12-102
Record Dates: First submitted 2013-05-03; First posted 2013-06-04 (Estimated); Results first posted 2016-11-11 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Pulmonary Disease
Keywords: Pleural Air Leak; Pulmonary resection; Video Assisted; Robotic Assisted
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Progel® Pleural Air Leak Sealant (Experimental)
  Interventions: Device: Progel® Pleural Air Leak Sealant

INTERVENTIONS:
Device: Progel® Pleural Air Leak Sealant — Video-assisted or robotic-assisted surgical lung procedures plus Progel® Pleural Air Leak Sealant

SUMMARY:
The objective of this clinical study is to evaluate the safety of the Progel® PALS, including the Progel® Extended Applicator Spray Tips, in sealing or reducing intraoperative air leaks in patients undergoing video assisted or robotic assisted thoracoscopic (VATS/Robotic) surgeries.

The data collected in this clinical study will supplement the Approved PMA P010047 Progel® PALS product.

DETAILED DESCRIPTION:
This is a prospective, open label, multi-center clinical study designed to assess the safety of the Progel® PALS product, including the Extended Applicator Spray Tip, when used in Video Assisted and Robotic Assisted Thoracoscopic Surgery. The study will treat approximately 105 evaluable subjects at up to 15 U.S. sites. All subjects will provide informed consent prior to enrollment in the study.

Patients who have met the initial screening criteria and who have a visible pleural air leak which requires treatment with a sealant, after standard closure techniques are used (standard sutures, staples or devices supplied by the hospital for thoracoscopic surgery) will be eligible for study participation. If the subject is treated, the surgeon will utilize Progel® PALS to the same sites originally treated with standard technique.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to provide written informed consent.
* Subject is scheduled for video assisted or robotic assisted thoracoscopic surgery for lung resection (i.e. lobectomy, bilobectomy, segmentectomy, and wedge resection/lung volume reduction), decortications or biopsy within 45 days of the screening evaluation.
* Subject is ≥18 years of age.
* Subject has a life expectancy ≥6 months.
* Following lung resection, subject has at least one or more visible intraoperative air leaks, after standard closure techniques are applied, that requires treatment with pleural sealant.
* Subject is willing and able to comply with the study procedures and complete the entire study as specified in the protocol, including the follow-up visits.

Exclusion Criteria:

* Subject has undergone previous lung resection or previous use of a sealant for air leaks.
* Subject has a serum creatinine ≥2.5 mg/dl at baseline or is currently on dialysis.
* Following lung resection, subject has intraoperative air leaks that require non-standard, visceral pleural closure (e.g. leak is too small or tissue is too fragile to use sutures/staples).
* Subject has any condition that, in the opinion of the Investigator, would preclude the use of the study device, or preclude the subject from completing the follow-up requirements.
* Subject has known allergy to human albumin or any component in the Progel® PALS product.
* Subject has an active or latent infection which is systemic or at the intended surgery site.
* Subject has necrotic or friable borders of the defect that will not support secure suture fixation if use of sutures is required.
* Subject is participating in another investigational drug or device trial.
* Subject is pregnant or has plans to become pregnant during the study period or is currently breastfeeding.
* Subject is part of the site personnel directly involved with this study.
* Subject is a family member of the investigational study staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Park, MD, Principal Investigator — Hackensack Meridian Health; John Snider, MD, Principal Investigator — Dean Foundation for Health, Research and Education, Inc
Locations (15):
- United States (15):
  - Cardiothoracic & Vascular Surgical Associates, PA, Jacksonville, Florida
  - Jupiter Medical Center, Inc., Jupiter, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute Hospital, Inc., Tampa, Florida
  - North Shore University Health System, Evanston, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Integrated Cardiology Group, LLC, Lincoln, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Trustees of Columbia University, NY - Presbyterian Hospital, New York, New York
  - Greenville Hospital System, Greenville, South Carolina
  - Baylor Research Institute, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - INOVA Health Care Services, Falls Church, Virginia
  - Dean Foundation for Health, Research, and Eduation, Inc, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park BJ, Snider JM, Bates NR, Cassivi SD, Jett GK, Sonett JR, Toloza EM. Prospective evaluation of biodegradable polymeric sealant for intraoperative air leaks. J Cardiothorac Surg. 2016 Dec 12;11(1):168. doi: 10.1186/s13019-016-0563-3. PMID 27955681

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in June 2013. 112 subjects were treated across 15 sites.
Pre-assignment Details: 207 subjects were consented and 112 were treated with Progel® PALS. Of the subjects who were not treated, 69 failed to meet intra-operative inclusion criteria (54/94 screened video-assisted subjects and 15/87 screened robotic assisted subjects) and 11 did not have a video or robotics procedure performed (ie, converted to open thoracotomy)
Period: Overall Study
Arm/Group | Progel® Pleural Air Leak Sealant
Started | 112
Completed | 103
Not Completed | 9
Not completed — Withdrawal by Subject | 6
Not completed — Death | 2
Not completed — Subject could not be contacted | 1

BASELINE CHARACTERISTICS:
Arm/Group | Progel® Pleural Air Leak Sealant
Number analyzed (Participants) | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 46
Region of Enrollment [Number; unit: participants]
  United States | 112

OUTCOME MEASURES:

1. Primary Outcome: Rate of Device and/or Procedure-related Adverse Events
Description: The primary outcome of the study is the rate of device- and/or procedure-related adverse events at one month after surgery in subjects using Progel® PALS in a VATS/Robotic procedure. Endpoint analysis of the rate of device- and/or procedure-related adverse events will be based on the Clinical Events Committee (CEC) adjudication of adverse events.
Time Frame: One (1) month follow-up
Population: Number of subjects reflects subjects who have completed 1-month follow-up visit or had device/procedure related AE before discontinuation.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Progel® Pleural Air Leak Sealant
Number analyzed (Participants) | 106
percentage of participants | 42.5 [34.3 to 50.9]

2. Secondary Outcome: Percentage of Subjects Without Postoperative Air Leaks Following Lung Surgery up to One (1) Month Follow-up
Time Frame: One (1) month
Population: MITT Population
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Progel® Pleural Air Leak Sealant
Number analyzed (Participants) | 112
percentage of participants | 49.1 [41.0 to 57.3]

3. Secondary Outcome: Percentage of Air Leaks That Are Sealed or Reduced
Time Frame: Day 0
Population: Subjects in the mITT population
Measure: Number (95% Confidence Interval); unit: percentage of air leaks
Units Other Than Participants: Number of Air Leaks
Arm/Group | Progel® Pleural Air Leak Sealant
Number analyzed (Participants) | 112
Number analyzed (Number of Air Leaks) | 133
percentage of air leaks | 96.2 [91.4 to 98.8]

4. Secondary Outcome: Number of Subjects Who Are Free From Air Leaks Immediately Following Surgery
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Progel® Pleural Air Leak Sealant
Number analyzed (Participants) | 112
Participants | 55

5. Secondary Outcome: Duration of Postoperative Air Leaks From the Time of Surgery Until the Air Leak Seals
Time Frame: Day 0-46
Population: MITT population minus 1 subject with missing data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Progel® Pleural Air Leak Sealant
Number analyzed (Participants) | 111
Days | 2.8 (6.75)

6. Secondary Outcome: Duration of Chest Tube Drainage
Time Frame: Day 0-46
Population: MITT Population minus 1 subject with missing data
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Progel® Pleural Air Leak Sealant
Number analyzed (Participants) | 111
Days | 4.3 (6.02)

7. Secondary Outcome: Duration of Hospitalization (Length of Stay)
Time Frame: Days 0-20
Population: MITT Population minus 2 subjects who died prior to discharge
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Progel® Pleural Air Leak Sealant
Number analyzed (Participants) | 110
Days | 4.6 (3.48)

8. Secondary Outcome: Patient Reported Quality of Life as Measured by the SF-36 at Change From Baseline at One(1) Month Follow up
Description: The scale ranges from 0 (minimum score) to 100 (maximum) score. A higher the score represents a more favorable health rating. The SF-36 was completed at baseline before surgery and one month post index procedure; the change calculation for both mental and physical components is based on the difference in scores between these two time points.
Time Frame: Baseline and One (1) Month Follow-up
Population: MITT Population minus 19 subjects with missing data at either baseline or 1 month post-procedure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Progel® Pleural Air Leak Sealant
Number analyzed (Participants) | 93
units on a scale
  Mental Component Score | -0.2 (9.20)
  Physical Component Score | -6.5 (9.98)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected through the one month follow-up period.
Arm/Group | Progel® Pleural Air Leak Sealant
Serious Adverse Events (participants affected / at risk) | 28/112
Other Adverse Events (participants affected / at risk) | 31/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Progel® Pleural Air Leak Sealant (N=112)
Cardiac Arrest (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Multi-organ Failure (General disorders) | 1
Pneumonia (Infections and infestations) | 3
Urinary Tract Infection (Infections and infestations) | 1
Post-procedural Hemorrhage (Injury, poisoning and procedural complications) | 1
Hyponaturemia (Metabolism and nutrition disorders) | 1
Carcinoid Tumor Pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Bronchial Secretion Retention (Respiratory, thoracic and mediastinal disorders) | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopleural Fistula (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneurmonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Air Leakage (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Progel® Pleural Air Leak Sealant (N=112)
Pyrexia (General disorders) | 12
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6
Arrythmia Supraventricular (Cardiac disorders) | 5
Pain (General disorders) | 3
Urinary Tract Infection (Infections and infestations) | 4
Mental Status Changes (Psychiatric disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary Air Leakage (Respiratory, thoracic and mediastinal disorders) | 3
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days